CLINICAL TRIAL: NCT01635075
Title: Acute Effects of Exercise in Smokers With Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brown University (Other)
Responsible Party: Principal Investigator, Jennifer Tidey, Associate Professor (Research), Brown University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 1R21DA031283 (NIH)
Record Dates: First submitted 2012-06-19; First posted 2012-07-06 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-09

CONDITIONS: Tobacco Dependence; Cigarette Craving; Smoking Behavior
Keywords: psychiatric; comorbidity; craving; tobacco
MeSH Terms: conditions — Tobacco Use Disorder; Smoking | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise (Experimental): 1-mile treadmill walk
  Interventions: Behavioral: Exercise
- Passive (Placebo Comparator): 20 min inactivity
  Interventions: Behavioral: passive control

INTERVENTIONS:
Behavioral: Exercise — 1-mile treadmill walk
  Arms: Exercise
Behavioral: passive control — 20 min inactivity
  Arms: Passive

SUMMARY:
People with schizophrenia have two- to three-times the mortality risk of the general population. This is primarily due to their unusually high rates of cigarette smoking, as well as other cardiovascular risk factors such as physical inactivity, obesity, high blood cholesterol and diabetes. Effective smoking treatments are needed to reduce morbidity and mortality in this population. Over a dozen experimental studies indicate that walking and other forms of exercise acutely reduce cigarette craving, nicotine withdrawal symptoms and smoking behavior in non-psychiatric smokers. However, the effects of acute exercise on smoking measures have not been studied in smokers with schizophrenia. This study will use a within-subjects, repeated-measures design, in which participants will undergo 4 laboratory sessions (order counterbalanced across participants): (1) smoking cues followed by exercise, (2) smoking cues followed by passive activity, (3) neutral cues followed by exercise, (4) neutral cues followed by passive activity. Outcome measures include cigarette craving, nicotine withdrawal symptoms, mood and smoking behavior. If the results of this study indicate that walking acutely reduces craving and smoking in smokers with schizophrenia, the next step in this research would be to test the effectiveness of a smoking cessation intervention that incorporates exercise bouts as a behavioral strategy for improving smoking cessation rates in this population.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of schizophrenia
* smoke at least 20 cigarettes per day
* less than 60 min moderate-intensity exercise per week

Exclusion Criteria:

* medication changes in past 4 weeks
* unable to give informed consent to participate
* alcohol/drug screen
* pregnant or nursing
* receiving or seeking immediate smoking treatment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-06; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Cigarette craving | within 10 minutes before and after exercise (or control activity)
  Questionnaire on Smoking Urges - Brief form

SECONDARY OUTCOMES:
Mood | within 10 minutes before and after exercise (or control activity)
  Positive and Negative Affect Scales, which are brief questionnaire measures of positive and negative mood.
Smoking habit withdrawal | within 10 minutes before and after exercise (or control activity)
  Questionnaire measures of withdrawal from sensorimotor aspects of smoking
Smoking choice | initiated 10 minutes after exercise (or control activity)
  2-hr laboratory smoking choice assessment in which participants make a series of choices between smoking versus receiving a small amount of cash.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Tidey, Ph.D., Principal Investigator — Brown University
Locations (1):
- Brown University, Providence, Rhode Island, United States

REFERENCES:
- See also: Research site — http://research.brown.edu/research/profile.php?id=1100925335